CLINICAL TRIAL: NCT04582474
Title: Demonstration of an Electronic Clinical Decision Support Module for Dengue Case Management and Reporting in Burkina Faso
Brief Title: Demonstration of an Electronic Clinical Decision Support Module for Dengue in Burkina Faso
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Ministry of Health, Burkina Faso (Other Government); Terre des hommes, Burkina Faso & Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FE008
Record Dates: First submitted 2020-09-08; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Dengue
Keywords: Non-malarial fevers; Clinical decision support tools; Rapid diagnostic test
MeSH Terms: conditions — Dengue | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dengue module and rapid diagnostic tests (Experimental)
  Interventions: Other: Dengue module and rapid diagnostic tests

INTERVENTIONS:
Other: Dengue module and rapid diagnostic tests — Digital platform providing clinical decision support for Dengue, Dengue rapid diagnostic tests and training will be deployed at study sites for Dengue screening, diagnosis, case management as well as reporting to surveillance system following local guidelines

SUMMARY:
The Integrated Management of Childhood Illness (IMCI) guideline has been implemented in Burkina Faso and is used across primary health facilities to assess children under the age of 5 years. A part from a rapid diagnostic test (RDT) for malaria, no other point of care in vitro diagnostic tests are widely used to improve disease diagnosis and inform treatment decisions. Dengue fever has been reported in Burkina Faso since 1925 and the recent epidemics in 2016 and 2017 have prompted the government to validate and deploy a clinical management algorithm for Dengue and a case reporting process to support surveillance for a targeted response.

The organisation Terre des hommes has digitalised IMCI and implemented the module through its Integrated electronic Diagnosis Approach (IeDA) programme across primary health care centers (PHCs) in the country with proven impact on clinical care and proven reduction in antibiotic prescriptions. Many recognize the need to update the IMCI guideline with current evidence. However this is challenging and may require large clinical trials. The advantage of electronic clinical decision support systems is plural: they improve quality of care through increased adherence and feedback information to the system; they strengthen surveillance systems by connecting relevant patient related data and provide geo-tagged coordinates for targeted responses; and they can become evidence-adaptive.

An electronic module of the Burkina Faso Dengue clinical management guideline accompanied with dengue rapid diagnostic tests has the potential to improve the diagnosis of non-malaria fevers in particular during "dengue seasons" and improve the efficiency of surveillance for this disease.

In this study, the investigators aim to assess the usability and the performance of the dengue module for patient management in primary health care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Older than 6 month
* Presentation with fever (axillary temperature ≥ 37,5⁰C) or history of fever for 2-7 days without localizing signs of another pathology such as malaria diagnosed by RDT
* Malaria diagnosis: negative malaria RDT performed at the the study site by a nurse as part of the routine consultation, or a positive malaria RDT with antimalarial treatment failure

Exclusion Criteria:

* Neonates (0-2 months) and children ≤ 6 month for operational reasons such as difficulties with blood draw
* Patients with severe disease requiring urgent care

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Point estimates of the percentage of dengue consultations performed using the dengue module, with 95% confidence intervals | 4 months
  This outcome will be evaluated by reporting the ratio of dengue consultations performed using the dengue module over the total number of consultations, together with a 95% confidence interval based on Wilson's score method.
Evaluation of the adherence to the different steps of the module | 4 months
  This outcome will be evaluated by the percentage ratio of dengue module steps adhered by patients over the total number of patients at each step.

SECONDARY OUTCOMES:
Estimate of the operational characteristic, Efficacy, of the dengue module: percentage of forms emitted from the module received in the surveillance system | 4 months
Estimate of the operational characteristic, Timeliness, of the dengue module: percentage of forms that are received by the surveillance system on time, as defined by the national surveillance system. | 4 months
Estimate of operational characteristic, Completeness, of the dengue module: percentage of fields that are completed. | 4 months
Positive predictive value of dengue rapid diagnostic test | 4 months
  Polymerase chain reaction results will be used as the reference test.

CONTACTS AND LOCATIONS:
Overall Officials: Brice W Bicaba, MD, Principal Investigator — Ministry of Health, Burkina Faso
Locations (2):
- Burkina Faso (2):
  - Centre de Santé et de Promotion Sociale (Sandogo), Ouagadougou, District Boulmiougou
  - Centre de Santé et de Promotion Sociale (Secteur 16), Ouagadougou, District Boulmiougou

IPD SHARING:
Plan to Share IPD: No